CLINICAL TRIAL: NCT02761525
Title: Topical Application of Silver Nanoparticles Reduced Oral Pathogens in Mechanically Ventilated Patients: A Randomized Controlled Clinical Trial
Brief Title: Topical Application of Silver Nanoparticles and Oral Pathogens in Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Francisco Javier Tejeda Nava, Dental Surgeon, Oral Pathology and Medicine, Clinical Profesor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UASLPFJTN
Record Dates: First submitted 2016-01-08; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Critical Illness
Keywords: silver nanoparticles antimicrobial activity
MeSH Terms: conditions — Critical Illness | interventions — colloidal silver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gel silver nanoparticles (Experimental): topic gel silver nanoparticles 12 ppm
  Interventions: Other: silver nanoparticles
- placebo (Placebo Comparator): topic innocuous gel
  Interventions: Other: placebo

INTERVENTIONS:
Other: silver nanoparticles — Allocation was randomized. Evaluate the effectiveness of silver nanoparticles incorporated into an innocuous gel and dished in oral mucosa surface to then compare with another innocuous gel without silver nanoparticles to reduce microbial colony forming units of pathogenic potential.
  Arms: gel silver nanoparticles
Other: placebo — Compare with another innocuous gel without silver nanoparticles to reduce microbial colony forming units of pathogenic potential using the same procedure to dished the gel.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether oral topic silver nanoparticles are effective to reduce potential pathogen microbial loads in mechanical ventilation patients.

DETAILED DESCRIPTION:
All patients were performed with oral hygiene as recommended by the clinical practice guidelines for the prevention, diagnosis and treatment of pneumonia associated with mechanical ventilation. After that, placed the treatment of an innocuous gel compound with 12ppm of silver nanoparticles or gel alone according to randomization. Then obtain and plant samples taken before the treatment 6 hours after. Comparing the results of the baseline sample with the final.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least 24 hrs application endotracheal tube and ventilator support were nasogastric tube ,in the ICU of Hospital Central "Dr. Ignacio Morones Prieto"
2. Patients with at least 24 hours of ICU admission.
3. Sedo - analgesia patients in a coma or induced coma.
4. Over 15 years old
5. Informed consent signed by a family member or legal guardian of the patient.

Exclusion Criteria:

1. The patient is not taking part in another study that cause conflict with the present test.
2. Patients who develop bronchiectasis , severe or massive hemoptysis , cystic fibrosis.
3. Patients with known sensitivity to silver.
4. Patients who had reported difficult intubation in the record.
5. Patients whose physical condition does not allow the completion of the oral examination, proper sampling or application of gel.
6. Pregnant women
7. Patients with oral mucositis

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Compare Colony Forming Units after the intervention. Unique dosis. | Comparison of microbial colony forming units at 6 hr of treatment with gel application
  Before oral hygiene in the intubated patient, it was taken with sterile swab, a saliva sample which was sown in dextrose Sabouraud agar and tryptone soya agar. 6 hours later, placement of the experimental gel, retook saliva sample with a sterile swab and they seeded in the same agars . Colony forming units were counted before and after the intervention using semi-automated colony counter .

IPD SHARING:
Plan to Share IPD: No
in process